CLINICAL TRIAL: NCT01895205
Title: A Randomized Comparative, Open-Label Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered by High Single Dose In-fusions or Red Blood Cell Transfusion in Women With Severe Postpartum Iron Deficiency Anaemia
Brief Title: Treatment of Women After Severe Postpartum Haemorrhage
Acronym: PP-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: BioStata (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP-02
Record Dates: First submitted 2013-06-26; First posted 2013-07-10 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Severe Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — iron isomaltoside 1000; Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron isomaltoside 1000 (Experimental): A single dose of 1500 mg iron isomaltoside 1000 is given. The dose is diluted in 100 ml 0.9% sodium chloride and given over approximately 15 min.
  Interventions: Drug: Iron isomaltoside 1000
- Red blood cell transfusion (Active Comparator): Allogenic RBC transfusion is dosed to trigger Hb:
  * Women with Hb 5.5 - 6.4 g/dL (3.5-3.9 mmol/L) will receive 2 units of RBC
  * Women with Hb 6.5 - 8.0 g/dL (4.0-5.0 mmol/L) will receive 1 unit of RBC
  Interventions: Drug: Red blood cell transfusion

INTERVENTIONS:
Drug: Iron isomaltoside 1000
  Other Names: Monofer®
  Arms: Iron isomaltoside 1000
Drug: Red blood cell transfusion
  Arms: Red blood cell transfusion

SUMMARY:
The primary purpose of this study is to get explorative information about IV high single dose infusion of iron isomaltoside 1000 compared to RBC transfusion in the treatment of severe PP-IDA evaluated as physical fatigue

ELIGIBILITY:
Inclusion Criteria:

1. PPH > 1000 mL
2. Hb ≥ 5.5 and ≤ 8.0 g/dL (≥ 3.5 and ≤ 5.0 mmol/L)
3. Willingness to participate and signed the informed consent form

Exclusion Criteria:

1. Women aged < 18 years
2. Multiple births
3. Peripartum RBC transfusion
4. Known iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemosiderosis)
5. Known hypersensitivity to parenteral iron or any excipients in the investigational drug products
6. Women with a history of active asthma within the last 5 years or a history of multiple allergies
7. Known decompensated liver cirrhosis and active hepatitis
8. Women with HELLP (Haemolysis Elevated Liver enzymes Low Platelet count) syndrome (defined according to "Dansk Selskab for Obstetrik og Gynækologi guidelines")
9. Active acute infection assessed by clinical judgement
10. Rheumatoid arthritis with symptoms or signs of active joint inflammation
11. History of anaemia caused by e. g. thalassemia, hypersplenism or haemolytic anaemia (known haematologic disorder other than iron deficiency)
12. Not able to read, speak and understand the Danish language
13. Participation in any other clinical study where the study drug has not passed 5 half-lives prior to the baseline
14. Any other medical condition that, in the opinion of Investigator, may cause the patient to be unsuitable for completion of the study or place the patient at potential risk from being in the study. For example, a malignancy, uncontrolled hypertension, unstable ischaemic heart disease or uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Physical Fatigue | From exposure to 12 weeks post-exposure

SECONDARY OUTCOMES:
Change in Hb concentration | From baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12
Change in p-ferritin | From baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12
Fatigue symptoms | from baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12
Postpartum depression | From week 1 to 3, 8 and 12
Breastfeeding | From exposure to 12 weeks post-exposure
Number of adverse drug reactions (ADRs) | From baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12
Change in p-iron | From baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12
Change in p-transferrin | From baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12
Change in transferrin saturation (TSAT) | From baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12
Change in reticulocyte count | From baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12
Change mean reticulocyte haemoglobin content (CHr) | From baseline to day 1, 2, 3, 4, 5, 6 and 7, week 3, 8 and 12

OTHER OUTCOMES:
Change in anaemia symptoms | From Baseline to week 12
Change in gastrointestinal symptoms | From Baseline to week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen, Denmark